CLINICAL TRIAL: NCT06559488
Title: Effects of Intravitreal Bevacizumab Intraoperatively in The Prevention of Early Recurrent Vitreous Hemorrhage Post-Vitrectomy in Diabetic Vitreous Hemorrhage
Brief Title: IVB for Post-vitrectomy Hemorrhage in Diabetic Eyes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Padjadjaran (Other)
Collaborators: Cicendo Eye Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OPHTH-202408.01
Record Dates: First submitted 2024-08-14; First posted 2024-08-19 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Diabetic Retinopathy; Vitreous Hemorrhage
Keywords: Diabetic vitreous hemorrhage; Intravitreal bevacizumab; Pars plana vitrectomy; Proliferative diabetic retinopathy; Recurrent vitreous hemorrhage
MeSH Terms: conditions — Diabetic Retinopathy; Vitreous Hemorrhage | interventions — Bevacizumab

STUDY DESIGN:
Intervention Model Description: A parallel group design was employed. Patients requiring vitrectomy for diabetic non-clearing vitreous hemorrhage (VH) were divided into two groups:
  Intervention Group: Underwent vitrectomy followed by an intravitreal injection of bevacizumab (1.25 mg/0.05 mL).
  Control Group: Underwent vitrectomy alone.
Who Masked: Outcomes Assessor
Masking Description: While it was not possible to mask participants and surgeons to the treatment allocation due to the nature of the surgical intervention, efforts were made to mask the outcome assessors. This involved:
  Centralized Data Collection: All data related to patient outcomes (visual acuity, VH grading, complications) were collected on standardized forms and sent to a central data management center.
  Coded Data Entry: Patient identification numbers were used instead of names to prevent bias.
  Masked Data Analysis: The statistician conducting the analysis was blinded to group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bevacizumab Intravitreal (Experimental): Ten patients underwent pars plana vitrectomy under local anesthesia. Vitrectomy used 3 23-gauge sclerotomies, triamcinolone for hyaloid cleaning, and hemostasis by elevated pressure, endo-diathermy, or laser. Panretinal laser applied to unlasered retina. Retina examined for tears or bleeding. IOP set at 20mmHg, sclerotomies sutured if needed. Post-vitrectomy, 1.25 mg bevacizumab injected via 30-gauge needle in superotemporal or inferotemporal pars plana.
  Interventions: Drug: Bevacizumab Injection [Avastin]; Procedure: Pars Plana Vitrectomy
- Control (Experimental): Eight patients underwent pars plana vitrectomy under local anesthesia. Vitrectomy used 3 23-gauge sclerotomies, triamcinolone for hyaloid cleaning, and hemostasis by elevated pressure, endo-diathermy, or laser. Panretinal laser applied to unlasered retina. Retina examined for tears or bleeding. IOP set at 20mmHg, sclerotomies sutured if needed.
  Interventions: Procedure: Pars Plana Vitrectomy

INTERVENTIONS:
Drug: Bevacizumab Injection [Avastin] — Intravitreal bevacizumab (1.25 mg/0.05 mL) was injected at the completion of vitrectomy surgery.
  Other Names: Pars Plana Vitrectomy
  Arms: Bevacizumab Intravitreal
Procedure: Pars Plana Vitrectomy — routine procedure of pars plana vitrectomy in vitreous hemorrhage for proliferative diabetic retinopathy patients

SUMMARY:
Recurrent vitreous hemorrhage following pars plana vitrectomy (PPV) for proliferative diabetic retinopathy remains a significant complication with reported incidence ranging from 11 to 75%. Early and late recurrences are associated with various factors, including residual blood, fibrovascular tissue, and neovascularization. Despite attempts to reduce this complication with therapies like anti-fibrinolytic agents, gas tamponade, and peripheral cryotherapy, the outcomes remain unsatisfactory.

DETAILED DESCRIPTION:
Recurrent vitreous hemorrhage following pars plana vitrectomy (PPV) for proliferative diabetic retinopathy remains a significant challenge with high incidence and negative impact on visual outcomes. Despite various treatments, intravitreal bevacizumab (IVB) has shown potential in reducing post-operative vitreous hemorrhage (PO-VH). This study aims to determine the efficacy and safety of intraoperative IVB in preventing PO-VH in patients undergoing vitrectomy for diabetic vitreous hemorrhage. This prospective, randomized controlled trial compared patients receiving intraoperative IVB to a control group. The primary outcome was PO-VH incidence at one month, with secondary outcomes including visual acuity change, time to VH clearance, and safety. Outcome assessors were masked to the study treatment. Data on demographics, medical history, visual acuity, VH grading, intraoperative findings, and postoperative complications will be collected. Statistical analysis compared PO-VH incidence and other outcomes between groups. This study will provide valuable evidence on the efficacy and safety of intraoperative IVB in preventing PO-VH, contributing to improved clinical practice and patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with spontaneous, non-clearing vitreous hemorrhage for at least one month as the initial vitrectomy indication for diabetic retinopathy.

Exclusion Criteria:

* Patients with tractional retinal detachment (ART)
* Patients with severe fibrovascular traction,
* Patients with intravitreal gas or silicone oil tamponade at the end of surgery
* Patients with other eye diseases besides diabetic vitreous hemorrhage
* Patients with history of intravitreal bevacizumab injection in the last 3 months before surgery
* Patients with other health condition includes uncontrolled hypertension, a history of coagulopathy
* Patients with inability to attend follow-up examinations for at least 1 month
* Patients taking anti-aggregation and anti-platelet medications with abnormal bleeding time (BT) and clotting time (CT)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Incidence and Severity of Vitreal Hemorrhage Post-Operative | Day 1, 7, and 30
  Calculation of incidence of Vitreal Hemorrhage Post Operative based on grading (Grade 0, Grade 1, Grade 2, Grade 3, Grade 4) between two groups; higher grades are related to worse outcomes

SECONDARY OUTCOMES:
Post operative visual Acuity, compared between groups | Day 1, 7, and 30
  Visual acuity measured with a Snellen chart was converted to logarithm of the minimum angle of resolution (logMAR) for statistical analysis. Snellen visual acuity of finger counting was categorized as log MAR 2.0, and hand motion as log MAR 3.0

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad Eko Prayogo, MD, Principal Investigator — Faculty of Medicine Universitas Padjadjaran
Locations (1):
- Cicendo Eye Hospital, Bandung, Jawab Barat, Indonesia